CLINICAL TRIAL: NCT03300843
Title: A Phase II Trial to Evaluate the Ability of a Dendritic Cell Vaccine to Immunize Melanoma or Epithelial Cancer Patients Against Defined Mutated Neoantigens Expressed by the Autologous Cancer
Brief Title: Ability of a Dendritic Cell Vaccine to Immunize Melanoma or Epithelial Cancer Patients Against Defined Mutated Neoantigens Expressed by the Autologous Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: slow accrual
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Steven Rosenberg, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 170177; 17-C-0177
Record Dates: First submitted 2017-10-03; First posted 2017-10-04 (Actual); Results first posted 2019-12-13 (Actual); Last update posted 2019-12-13 (Actual); Status verified 2019-11

CONDITIONS: Melanoma; Gastrointestinal Cancer; Breast Cancer; Ovarian Cancer; Pancreatic Cancer
Keywords: Cell Therapy; Immunotherapy; Vaccines
MeSH Terms: conditions — Melanoma; Gastrointestinal Neoplasms; Breast Neoplasms; Ovarian Neoplasms; Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Peptide loaded dendritic cell vaccine (Experimental): Peptide loaded dendritic cell vaccine on days 0, 14, 28, and 42
  Interventions: Biological: Peptide loaded dendritic cell vaccine

INTERVENTIONS:
Biological: Peptide loaded dendritic cell vaccine — On days 0, 14 (+/- 5 days), 28 (+/- 5 days), and 42 (+/- 5 days). The vaccine will be administered as both an intravenous (IV) infusion and a subcutaneous (SQ) injection. The total dose will be divided equally between intravenous (IV) and SQ containing 1.0E7 to 8.0E7 cells per cycle depending upon the manufacturing yield.

SUMMARY:
Background:

Exomes are the parts of deoxyribonucleic acid (DNA) that make proteins. Researchers are finding a way to read the letters in the exome. Incorrect letters are called mutations. Tumors contain specific mutations. Researchers can find these mutations in tumors to make treatments. Researchers want to use pieces of participants tumors to find the tumor-specific mutations. They also will take participants white blood cells to make a vaccine that they hope will shrink the tumors.

Objectives:

To see if dendritic vaccine tumor-fighting cells are safe and can cause certain cancer tumors to shrink.

Eligibility:

Adults ages 18-70 who have metastatic melanoma or metastatic epithelial cancer

Design:

The first part of this study was done under protocol 03-C-0277. In that study, white blood cells and pieces of participants' tumors were taken to make a vaccine.

In this study, participants will get a vaccine every 2 weeks for 8 weeks. It will be given both in a vein and under the skin. At each visit, participants will have a physical exam and have blood taken. They will talk about any side effects they have.

After treatment ends, participants will have many follow-up visits for the first year, then once each year after that. Visits will last up to 2 days each. They will include lab tests, imaging studies, and a physical exam. Blood will be taken at each visit. At the first follow-up visit, participants may have leukapheresis, which they also had as part of protocol 03-C-0277. Participants may not have to return to the Clinical Center for these visits.

DETAILED DESCRIPTION:
Background:

* Therapeutic vaccination against cancer has proven very challenging with little clinical benefit.
* Vaccines against non-viral tumors have mainly targeted differentiation antigens, cancer testis antigens, and overexpressed antigens. However negative selection in the thymus against these normal nonmutated antigens severely limits the ability to generate high avidity anti-cancer T cells. Such depletion can impair their antitumor activity and limit tumor elimination.
* The National Cancer Institute Surgery Branch (NCI SB) has developed a pipeline for the identification of immunogenic T cell epitopes derived from neoantigens.
* In recent studies, we identified the neoantigens recognized by tumor infiltrating lymphocytes (TIL) that mediated regression in patients with metastatic cancer. Using whole exome sequencing of a resected metastatic nodule followed by high throughput immunologic screening, we were able to demonstrate that tumor regressions were associated with the recognition by the administered TIL of unique somatic mutations that occurred in the cancer.
* We, therefore, aim to use this pipeline to identify immunogenic neoantigens from epithelial cancer patients and to use these defined epitopes for a personalized therapeutic dendritic cell (DC) vaccine.

Objectives:

-Primary objectives:

--To determine the clinical response rate in patients with metastatic melanoma or epithelial cancer who receive this DC vaccine

Eligibility:

* Age greater than or equal to 18 and less than or equal to 70 years
* Eastern Cooperative Oncology Group (ECOG) 0 - 2
* Evaluable metastatic melanoma or epithelial cancer refractory to standard treatment
* Metastatic melanoma or epithelial cancer lesion(s) that is resectable for TIL or in selected cases, available peripheral blood mononuclear cells (PBMC).

Design:

* Patients with metastatic melanoma or epithelial cancer will undergo surgical resection of tumor followed by exome and ribonucleic acid (RNA) sequencing to identify expressed mutations (CONDUCTED UNDER THE National Cancer Institute Surgery Branch (NCI SB) COMPANION PROTOCOL 03-c-0277).
* Patients will undergo apheresis and DC will be cryopreserved for vaccine preparation.
* Immunogenic neoantigens will be identified from TIL and PBMC by high throughput immunologic screening using long peptides and tandem minigenes covering all mutated epitopes.
* Patient will be vaccinated with autologous mature dendritic cells loaded with long peptides and minimal epitopes from defined neoantigens or highly expressed mutations in tumor suppressor or driver genes.
* DC will be administered intravenously and subcutaneously for four cycles at biweekly intervals.
* Blood samples will be taken every two weeks, and patients will be monitored for the quantity and quality of circulating neoantigen-specific T cells.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Metastatic melanoma or epithelial cancer with at least one lesion that is resectable or in selected cases, available peripheral blood mononuclear cells (PBMCs)
* Measurable and evaluable metastatic disease per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria
* Confirmation of the diagnosis of metastatic cancer by the Laboratory of Pathology of National Cancer Institute (NCI).
* All patients must be refractory to approved standard systemic therapy.
* Patients with 3 or fewer brain metastases that are less than 1 cm in diameter and asymptomatic are eligible. Lesions that have been treated with stereotactic radiosurgery must be clinically stable for one month after treatment for the patient to be eligible. Patients with surgically resected brain metastases are eligible.
* Greater than or equal to 18 years of age and less than or equal to 70 years of age.
* Clinical performance status of Eastern Cooperative Oncology Group (ECOG) 0, 1, 2
* Patients of both genders must be willing to practice birth control from the time of enrollment on this study and for up to four months after treatment.
* Serology:

  * Seronegative for Human Immunodeficiency Virus (HIV) antibody. (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who are HIV seropositive can have decreased immune-competence and thus are less responsive to the experimental treatment and more susceptible to its toxicities.)
  * Seronegative for hepatitis B antigen, and seronegative for hepatitis C antibody. If hepatitis C antibody test is positive, then the patient must be tested for the presence of antigen by reverse transcriptase polymerase chain reaction (RT-PCR) and be hepatitis C virus ribonucleic acid (HCV RNA) negative.
* Hematology

  * Absolute neutrophil count greater than 1000/mm^3 without the support of filgrastim
  * White blood cell (WBC) greater than or equal to 3000/mm^3
  * Platelet count greater than or equal to 100,000/mm^3
  * Hemoglobin > 8.0 g/dl. Subjects may be transfused to reach this cut-off.
  * Cluster of differentiation 4 (CD4) count > 200/uL
* Chemistry:

  * Serum alanine aminotransferase (ALT)/aspartate aminotransferase (AST) less than 5.0 x ULN
  * Serum Creatinine less than or equal to 1.6 mg/dl
  * Total bilirubin less than or equal to 2.0 mg/dl, except in patients with Gilbert's Syndrome, who must have a total bilirubin less than or equal to 3.0 mg/dl.
* More than four weeks must have elapsed since any prior systemic therapy at the time the patient receives the vaccine, and patients toxicities must have recovered to a grade 1 or less (except for toxicities such as alopecia or vitiligo).

Note: Patients may have undergone minor surgical procedures within the past 3 weeks, as long as all toxicities have recovered to grade 1 or less.

* Ability of subject to understand and the willingness to sign a written informed consent document.
* Subjects must be co-enrolled On protocol 03-C-0277.

EXCLUSION CRITERIA:

* Women of child-bearing potential who are pregnant or breastfeeding because of the potentially dangerous effects of the treatment on the fetus or infant.
* Any form of primary immunodeficiency (such as Severe Combined Immunodeficiency Disease).
* Concurrent opportunistic infections (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who have decreased immune competence may be less responsive to the experimental treatment and more susceptible to its toxicities).
* Active systemic infections (requiring anti-infective treatment), coagulation disorders or any other active or uncompensated major medical illnesses.
* Patients who are receiving any other investigational agents.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2018-04-11 (Actual); Primary Completion 2019-07-09 (Actual); Study Completion 2019-09-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven A Rosenberg, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Klein L, Hinterberger M, Wirnsberger G, Kyewski B. Antigen presentation in the thymus for positive selection and central tolerance induction. Nat Rev Immunol. 2009 Dec;9(12):833-44. doi: 10.1038/nri2669. PMID 19935803
- [Background] Abramson J, Giraud M, Benoist C, Mathis D. Aire's partners in the molecular control of immunological tolerance. Cell. 2010 Jan 8;140(1):123-35. doi: 10.1016/j.cell.2009.12.030. PMID 20085707
- [Background] Bos R, Marquardt KL, Cheung J, Sherman LA. Functional differences between low- and high-affinity CD8(+) T cells in the tumor environment. Oncoimmunology. 2012 Nov 1;1(8):1239-1247. doi: 10.4161/onci.21285. PMID 23243587

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Peptide Loaded Dendritic Cell Vaccine
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Peptide Loaded Dendritic Cell Vaccine
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Who Had a Clinical Response (Complete Response (CR) + Partial Response (PR)) to Treatment
Description: Response was assessed by the RECIST v1.1. Complete Response is disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Partial Response is at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum of diameters.
Time Frame: up to 6 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Peptide Loaded Dendritic Cell Vaccine
Number analyzed (Participants) | 1
percentage of participants | 0

2. Secondary Outcome: Number of Participants With 2-3 Fold Increase From Baseline in Reactivity to Circulating Antigen-specific T Cells to the Mutated Peptide Compared to the Non-mutated Peptide
Description: Enzyme-linked immunosorbent assay (ELISA) and enzyme-linked immune absorbent spot (ELISpot) assays assessed reactivity to the mutated peptide compared to the non-mutated peptide. Differences of 2-3 fold in these assays over the baseline measurement are indicative of true biologic differences.
Time Frame: Day 0, Day 14 (± 5 d), Day 28 (± 5 d), and Day 42 (± 5 d)
Measure: Count of Participants; unit: Participants
Arm/Group | Peptide Loaded Dendritic Cell Vaccine
Number analyzed (Participants) | 1
Participants
  Mutated peptide Day 0 | 0
  Mutated peptide Day 14 | 0
  Mutated peptide Day 28 | 0
  Mutated peptide Day 42 | 0
  Non-Mutated peptide Day 0 | 0
  Non-Mutated peptide Day 14 | 0
  Non-Mutated peptide Day 28 | 0
  Non-Mutated peptide Day 56 | 0

3. Secondary Outcome: Number of Participants With Serious and Non-serious Adverse Events
Description: Here is the count of participants with serious and non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approximately 6 months and 11 days
Measure: Count of Participants; unit: Participants
Arm/Group | Peptide Loaded Dendritic Cell Vaccine
Number analyzed (Participants) | 1
Participants | 1

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 6 months and 11 days.
Arm/Group | Peptide Loaded Dendritic Cell Vaccine
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Peptide Loaded Dendritic Cell Vaccine (N=1)
Nausea (Gastrointestinal disorders) | 1 (4)
Fatigue (General disorders) | 1 (1)
Injection site reaction (General disorders) | 1 (6)
Headache (Nervous system disorders) | 1 (7)
Skin induration (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-03-26): https://cdn.clinicaltrials.gov/large-docs/43/NCT03300843/Prot_SAP_000.pdf
  • Informed Consent Form (2018-04-04): https://cdn.clinicaltrials.gov/large-docs/43/NCT03300843/ICF_001.pdf